CLINICAL TRIAL: NCT05913063
Title: Direct Discrimination of Quantum States by the Human Eye With Macular Degeneration
Brief Title: Direct Discrimination of Quantum States by the Human Eye
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Eye and Vision Research (Other)
Collaborators: University of Waterloo (Other); The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SLIM
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-Related Macular Degeneration; Structured Light; Orbital Angular Momentum; Polarization Perception; Retinal Imaging
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Within-subject, measuring the threshold SL-based entoptic phenomenon circular obstruction size of the radial retinal polarizer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Age-Related Macular Degeneration (Experimental): Conducting the psychophysical task on the perception of OAM-coupled polarized light
  Interventions: Device: Structured Light Imaging Microscopy

INTERVENTIONS:
Device: Structured Light Imaging Microscopy — Conducting the psychophysical task on the perception of OAM-coupled polarized light created using the experimental setup - Structured Light Imaging Microscopy (SLIM). Four types of vortex orbital angular momentum, differing by the number of fringes l=5;10; 15;20, will be presented for 0.5s per trial during which an azimuthally varying entoptic profile rotated clockwise or counterclockwise. A circular mask with a varying radius will be placed at fixation, thus the task will be performed at varying eccentricities. Circular obstruction of the area will be achieved due to the high refresh-rate structured light modulator. The threshold mask size will be changed by a 2up/1down staircase method (71% accuracy for the estimation of mask size).

SUMMARY:
Age-related macular degeneration (AMD), is a debilitating eye disease that causes a loss of central vision. The prevalence of AMD increases exponentially with age and causes a significant impact through both medical expenses and the social and economic costs associated with vision loss. AMD is the global leading cause of blindness among people over the age of 60. Detection of this eye disease at early stages coupled with prompt treatment can prevent vision loss; however, modern diagnosis methods are ineffective at diagnosis of AMD before vision loss occurs. While a range of available treatment options has been effective at slowing vision loss due to AMD, no treatment exists which can recover lost vision. The investigators propose to apply tools developed in quantum information science to diagnose AMD before vision has been affected, drastically improving health outcomes for patients with AMD.

DETAILED DESCRIPTION:
There has been tremendous progress in generating and detecting structured light which possesses advantageous propagation characteristics such as quantized orbital angular momentum (OAM), non-diffraction, and self-healing. These special beams have found applications in microscopy, encoding and multiplexing of communications, and manipulation of matter. Here the investigators bring the structured light toolbox to vision sciences for the first time and expand the space of possible stimuli.

A healthy macula possesses azimuthally ordered dichroic fibres that act as a radial polarization filter, enabling a typical person to perceive linearly polarized light through the entoptic phenomena known as Haidinger's brushes. Despite significant interest in the application of this phenomenon to the detection of age-related macular degeneration, no device has currently seen widespread adoption in a clinical environment. This is due to the difficulty in observing Haidinger's brush, the imprecise measurements that this test can extract, and the difficulty in instructing patients during these tests.

Leveraging the quantum-inspired toolbox developed in the field of structured light, the investigators can project polarization-coupled OAM states of light directly on a person's retina. This enables the investigators to create arbitrary entoptic patterns in a person's vision based on the structure and chemical composition of their subjective macula, and the investigators have the opportunity to develop a litany of novel diagnostic tests to characterize and quantify the health of the macula.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are clinically diagnosed with a vision disease affecting their macula
* Older adults who are matched for age.
* Participants who are clinically diagnosed with glaucoma
* Participants who have normal vision.
* One aged-matched control with normal vision will be recruited for each of the diagnosed groups (born in the same year).

Exclusion Criteria:

* Participants with any additional eye diagnosis or condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Perception of the structured light | Approximately 10 minutes, Screening and Training day (Session 1)
  Assessment of the participant's ability to see the entoptic phenomena created using the structured light (SL) - orbital angular momentum (OAM) coupled polarized light. Various SL vortex and radial patterns will be projected using the custom research-based laser optical setup
Radius of the radial retinal polarizer | Approximately 30 minutes, on the completion of the study (Session 6)
  Calculation of the radius of the central obstruction. From a total of 14 reversal trials, the six last values of the mask size will be used for the calculation of the threshold mask size mean (r mean). The standard deviation will be computed from the variance of these last six trials

SECONDARY OUTCOMES:
Thickness of retina and retinal layers | Approximately 10 minutes, Screening and Training day (Session 1)
  Measurement of the retinal layers' thickness and total neuroretina
Contrast sensitivity | Approximately 5 minutes, Screening and Training day (Session 1)
  Computer-based measurement of contrast sensitivity
Fundus photography | Approximately 5 minutes, Screening and Training day (Session 1)
  Imaging the retina using white light. The diameter of the optic nerve head will be measured in order to calculate the degree/pixel ratio for each participant
Ocular biometry measurement | Approximately 5 minutes, Screening and Training day (Session 1)
  Measurement of the central corneal thickness and axial eye length
Macular pigment optical density measurement | Approximately 10 minutes, Screening and Training day (Sessions 1 and 2)
  Computer-based measurement of the macular pigment optical density (MPOD)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Thompson, PhD, Principal Investigator — Centre for Eye and Vision Research; Mukhit Kulmaganbetov, MD, PhD, Study Director — Centre for Eye and Vision Research
Locations (1):
- Centre for Eye and Vision Research Limited, Hong Kong, Guangdong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared on request
Supporting Information: Study Protocol
Time Frame: After the publication of study results for an indefinite period.
Access Criteria: Upon reasonable request and approved by the study principal investigator.